CLINICAL TRIAL: NCT04862000
Title: Prospective Long Term Observational Study of Health Profile, Clinical Characteristics and Outcome of Patients Suffering From Endometriosis and Adenomyosis
Brief Title: Observational Study of Patients Suffering From Endometriosis and Adenomyosis
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Fung Wen Ying Linda, Associate Consultant, Chinese University of Hong Kong
Other Study IDs: CRE 2020.688
Record Dates: First submitted 2021-03-27; First posted 2021-04-27 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Endometriosis; Adenomyosis
Keywords: Endometriosis; Adenomyosis
MeSH Terms: conditions — Endometriosis; Adenomyosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Endometriosis or adenomyosis: participants suffering pelvic endometriosis, endometrioma, deep infiltrating endometriosis or adenomyosis

SUMMARY:
Endometriosis and adenomyosis are chronic difficult diseases affecting a significant proportion of reproductive age women. it is hoped that the investigators can collect the health profile of these participants using structured questionnaires on their quality of life, reproductive health, collect the sonographic characteristics, identify the risks factors of participants suffering from severe disease, and to propose the best treatment modality for different patient groups, both with and without fertility wish.

DETAILED DESCRIPTION:
Endometriosis and adenomyosis are chronic difficult diseases affecting a significant proportion of reproductive age women. Not only the disease can lead to chronic pelvic pain, dyspareunia and dysmenorrhea, it is also associated with impaired reproductive health, infertility and tubal-peritoneal disease. Adenomyosis can also result in anaemia due to the increased uterine volume and menstrual blood loss. Different treatment options are available for this group of participants, ranging from simple medical treatment to control symptoms, such as analgesics for pain control, transexemic acid to reduce menstrual blood loss, to hormonal treatment and the more radical surgical treatment.

As a tertiary gynaecology referral centre, the investigators encounter a large volume of patients suffering from endometriosis and adenomyosis of different disease severity. Through this prospective observational study, it is hoped that the investigators can collect the health profile of participants using structured questionnaires on their quality of life, reproductive health, collect the sonographic characteristics, identify the risks factors of patients suffering from severe disease, and to propose the best treatment modality for different participant groups, both with and without fertility wish.

Patients attending the pelvic mass clinic/ endometriosis clinic with the histologically confirmed or sonographic evidence of endometriosis/ adenomyosis will be invited to participate in the prospective study. Their demographic data will be collected. Symptomatology and health profile will be collected via questionnaires (e.g.EHP-30, SF 36, FSFI) to evaluate the physical, psychological, sexual and social aspects of patients affecting by the disease. Menstrual chart with be recorded. Physical examination including abdominal and pelvic examination will be performed. Pelvic sonography will be offered and recorded systematically. Different medical/ surgical treatments will be offered based on patient's clinical condition in an evidence-based approach and clinical guidance. Their treatment outcome will be assessed during the follow-up. Surgical findings will be recorded and disease severity graded by use of AFS scores. Pathological findings will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* with endometriosis or adenomyosis confirmed by ultrasound or MRI

Exclusion Criteria:

* refuse to participate in the study, less than 18 years old, menopausal, illiterate or mentally incapable

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Patients with endometriosis or adenomyosis treated in the Department of Obstetrics and Gynaecology, Prince of Wales Hospital, Shatin, Hong Kong
Sampling Method: Probability Sample
Enrollment: 880 (Estimated)
Dates: Start 2021-04-30 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Endometriosis Health Profile (EHP-30) questionnaire score | from enrollment to end of treatment at five years.
  The Endometriosis Health Profile-30 (EHP-30) is a disease-specific questionnaire to measure the health-related quality of life in patients with endometriosis. EHP-30 score is ranging from 0 (best health status) to 100 (worst health status). EHP-30 questionnaire score before and after medical and surgical treatment will be evaluated.
Visual Analog Scale (VAS) pain score | from enrollment to end of treatment at five years.
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by participant making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain." Mean change in pain score on VAS before and after medical and surgical treatment will be evaluated.

SECONDARY OUTCOMES:
side effects profile of medical treatment | from the first follow up at six months to end of treatment at five years.
  side effects profile of medical treatment for endometriosis and adenomyosis. The bone mineral density measurement (DEXA) will be arranged if participants has prolonged usage of progestogens over 2 years. Menstrual pattern will be recorded using menstrual calendar.
ultrasound findings correlation with surgical findings | from enrollment to three months post-surgery
  ultrasound findings correlation with surgical findings using AFS scores and Endometriosis fertility index EFI scores
symptoms recurrence | from enrollment to end of treatment at five years.
  symptoms recurrence including pelvic pain, menstrual problems and endometrioma recurrence after medical or surgical treatments
reproductive outcome | from enrollment to end of treatment at five years.
  evaluate the reproductive outcome in those participants with fertility wish. Spontaneous pregnancy rates and requirement for assisted reproductive technology after surgery will be studied, with reference to the intraoperative AFS scores.

CONTACTS AND LOCATIONS:
Overall Officials: Wen Ying Linda FUNG, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No